CLINICAL TRIAL: NCT07250893
Title: Resolving Early Life Stress: Psychotherapy Outcomes and Neurobiology in Complex Depression
Acronym: RESPOND
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Sun Life Financial Movement Disorders Research and Rehabilitation Centre (Other)
Responsible Party: Principal Investigator, Benicio Frey, Professor, Psychiatry & Behavioural Neurosciences; Director, Women's Health Concerns Clinic, St. Joseph's Healthcare Hamilton, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17671
Record Dates: First submitted 2025-04-08; First posted 2025-11-26 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Depression - Major Depressive Disorder; Childhood Traumas
Keywords: Early life adversity; Depression; Emotional dysregulation; Childhood trauma
MeSH Terms: conditions — Depression | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychotherapy arm (Experimental): The psychotherapy intervention will be delivered virtually over 12 weeks, 1x/week for 1 hour, 1-on-1 with a therapist
  Interventions: Other: Psychotherapy

INTERVENTIONS:
Other: Psychotherapy — Session 1 - Psychoeducation: Introductions + information about adversity and depression
  Session 2 - Behavioural Activation: Identify activation targets, create Daily Activities Schedule
  Session 3 - Identifying Emotions: Describe + label emotions; cycle of emotions
  Session 4 - Distress Tolerance: STOP + TIP skills
  Session 5 - Distress Tolerance: Self-soothing + improving the moment
  Session 6 - Stuck Points: Stuck points + impact statements
  Session 7 - Self-blame Beliefs: Negative self schemas; alternative thoughts worksheet
  Session 8 - Safety + Trust: Schemas of emotional safety and trust about self and others
  Session 9 - Power + Control: Stuck points related to scope of influence over events + the world
  Session 10 - Esteem: Reconstruct ideas of self; engaging positively with others
  Session 11 - Intimacy: Develop self- and other intimacy behaviours
  Session 12 - Wrap-up: Review new impact statements; revisit behavioural chang

SUMMARY:
The RESPOND trial explores the link between early life adversity and later life depressive symptoms. The investigators have designed a new psychological therapy tailored to address the symptoms that can be caused by difficult experiences in early life. These symptoms include low mood, emotional dysregulation, and distressing thoughts and beliefs related to difficult or traumatic experiences. The investigators would like to see if this new therapy helps people feel better. The investigators are also studying the biological changes that can occur as a result of early life adversity, and how this therapy may influence those changes. To do this, the investigators ask questions about participants' physical and mental health and take blood samples.

DETAILED DESCRIPTION:
Objectives of proposed study:

1. Assess efficacy of a novel psychotherapy protocol:

   The investigators will evaluate a new psychotherapy specifically designed to target depressive symptoms and emotional dysregulation in individuals with depressive symptoms and a history of ELA. This protocol incorporates evidence-based techniques from Dialectical Behavior Therapy (DBT), Cognitive Behavioral Therapy (CBT), and Cognitive Processing Therapy (CPT), and is tailored to the unique needs of this population.
2. Examine biological mechanisms underlying the link between ELA and depression:

To investigate the biological processes that link ELA to later-life depressive pathology, the study will explore epigenetic, inflammatory, and hormonal markers, as well as clinical mechanisms such as trauma-related factors, illness presentation, and comorbid diagnoses.

The primary outcome of this study is a change in depression symptoms as characterized by the Montgomery Åsberg Depression Rating Scale (MADRS). The secondary outcomes will be changes in emotional regulation as measured by the Difficulties in Emotional Regulation Scale (DERS), changes in trauma symptoms as measured by the PTSD Checklist for the DSM-5 (PCL-5) and the International Trauma Questionnaire (ITQ), and changes in inflammation and methylation status as measured through blood analysis.

This study will be run as an open-label, single arm, proof of concept intervention study. The intervention will be run in virtually, 1-on-1, 1x/week for 12 weeks. Participants will undergo a baseline assessment before treatment begins, including biological and clinical measurements; during treatment weekly measures will be administered using the myCap application; more extensive clinical assessments will be done at treatment midpoint (treatment week 6); biological and clinical measurements will be collected at treatment end point (treatment week 12); clinical measures will be collected at a follow-up timepoint (3 months post-treatment).

This study will enroll assigned female at birth (18+) participants with depressive symptoms as measured by the Hamilton Depression Rating Scale (HAM-D) and history of early adversity as indicated by the Childhood Experiences of Care and Abuse questionnaire (CECA q) or the Adverse Childhood Experiences questionnaire (ACES q).

Inclusion:

* Adults 18 years old or older
* at or over 18 on HAM-D, indicative of moderate-severe depressive symptoms
* Any childhood (before 18 years old) adversity as indicated by scores on the CECA q and ACES q

The broad inclusion criteria were chosen in an effort to ensure the study captures a representative sample of people who experience depressive symptoms as a result of early life adversity. The investigators anticipate that some participants will meet criteria for a DSM-5 diagnosis of PTSD or ICD-11 diagnosis of PTSD or complex PTSD, but others will not. This study design will facilitate comparison of participants who develop threshold stress-related disorder symptoms against those who don't on clinical and biological measures, and impairment.

Exclusion:

* Individuals who meet for PTSD diagnosis from a criterion A trauma occurring in adulthood without a history of ELA

  o Individuals meeting DSM-5 PTSD criteria will be able to get appropriate care through trauma-focused clinics and treatments. Best-evidence treatment for PTSD is a better option for those who meet for a PTSD diagnosis from a criterion A trauma in adulthood (CPT, EMDR, etc.). Additionally, those with criterion A trauma from adulthood may not resonate with the components of the proposed psychotherapy.
* Individuals experiencing active mania or psychosis
* Individuals with an active substance use disorder
* Individuals presenting with active suicide risk (plan, intention, means) indicative of a need for higher level care
* Individuals in current psychotherapeutic treatment (defined as having engaged in consistent psychotherapy within the last 3 months)

Participants will attend in 4 visits outside of the treatment schedule:

* Screening visit

  * Can be done either in person or virtually
  * Consent obtained, eligibility assessed and confirmed
  * Information given about structure and content of psychotherapy
* Baseline visit

  * Must be done in person
  * Diagnostic interview done, blood collected, demographics and medical information collected, and clinical measures administered
* Treatment endpoint visit (Week 12)

  * Must be done in person
  * Blood collected and clinical measures administered
* Follow-up appointments

  * Can be done either in person or virtually
  * Clinical measures administered

The psychotherapy intervention was designed by Dr. Sheryl Green, Dr. Jenna Boyd, Dr. Francisco Lima, and Katerina Dikaios. Dr. Sheryl Green is a senior psychologist in the Women's Health Concerns Clinic, a fellow of the Canadian Association of Cognitive and Behavioural Therapies, and has successfully developed multiple novel cognitive behavioural therapy (CBT)-based interventions. Dr. Jenna Boyd is a senior psychologist in the Anxiety Treatment and Research Clinic and an expert in treating specific trauma populations with cognitive behavioural therapy modalities. Dr. Francisco Lima is a psychiatrist in the Women's Health Concerns Clinic, an experienced psychotherapist, and an expert in PTSD and complex trauma. Katerina Dikaios is a PhD candidate in the Psychology Research and Clinical Training program at McMaster University, under the supervision of Drs. Benicio Frey and Sheryl Green; she has an extensive background in psychiatric research including trauma assessment and depression treatment and is currently receiving comprehensive clinical training in cognitive behavioural therapies.

The rationale for this psychotherapy protocol is based on existing evidence suggesting that psychotherapies that prioritize emotional regulation skills before trauma focused therapy appear to garner positive results for individuals who have experienced complex trauma. To date, there has been no investigation of this strategy in individuals with depression. Because complex trauma frequently precedes depressive illness, we have identified this population as an important target for specific psychotherapeutic intervention.

The psychotherapy protocol integrates components from cognitive behavioural therapy (CBT), dialectical behavioural therapy (DBT), and cognitive processing therapy (CPT). The protocol was designed to address common clinical features previously identified in this population, namely low mood, emotional dysregulation, and stuck points related to trauma-related beliefs about oneself and the world. These features map on to ICD-11 cPTSD DSO symptoms clusters of emotional dysregulation (including low mood), negative self-concept, and disturbances in relationships.

Because existing literature has not explored treatment of complex trauma in the context of depressive illness, we tailored this treatment to the population by including aspects of CBT for depression (psychoeducation and behavioural activation) to provide participants with skills to aid in initial alleviation of depressive symptoms. CBT skills is followed by DBT skills hand selected to be applicable for emotional regulation difficulties in this population, along with cognitive processing therapy (CPT) techniques for targeted treatment of trauma-related symptoms.

The psychotherapy intervention will be delivered virtually over 12 weeks, 1x/week for 1 hours, 1-on-1 with a trained therapist. Virtual participation will be held over St. Joe's institutionally licensed Zoom or Teams account.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years old or older
* At or above 18 on HAM-D, indicative of moderate-severe depressive symptoms
* Any childhood (before 18 years old) adversity as indicated by scores on the CECA q and ACES q

Exclusion Criteria:

* Individuals who meet for PTSD diagnosis from a criterion A trauma occurring in adulthood without a history of ELA
* Individuals experiencing active mania or psychosis
* Individuals with an active substance use disorder
* Individuals presenting with active suicide risk (plan, intention, means) indicative of a need for higher level care
* Individuals in current psychotherapeutic treatment (defined as having engaged in consistent psychotherapy within the last 3 months)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2028-08-15 (Estimated)

PRIMARY OUTCOMES:
Montgomery and Asberg Depression Rating Scale (MADRS) | Baseline (week 0), Treatment endpoint (week 12), Follow-up (3 months post treatment)
  The Montgomery and Asberg Depression Rating Scale is a 10-item semi-structured interview assessing the severity of depressive symptoms (Montgomery & Åsberg, 1979). The MADRS is sensitive to changes induced my treatment, making it appropriate to implement over psychotherapeutic intervention to monitor changes in depression severity.

SECONDARY OUTCOMES:
Difficulties with Emotional Regulation Scale | Baseline (week 0), Treatment endpoint (week 12), Follow-up (3 months post treatment)
  The Difficulties with Emotional Regulation Scale is a self-report measure used to assess emotional regulation difficulties over multiple domains (Gratz & Roemer, 2004). It is a transdiagnostic measure appropriate for measuring changes in emotional regulation over time.
International Trauma Questionnaire | Baseline (week 0), Treatment endpoint (week 12), Follow-up (3 months post treatment)
  The International Trauma Questionnaire is a self-report measure designed to assess and diagnose PTSD and complex PTSD in accordance with criteria from the ICD-11 (Cloitre, 2020; Cloitre et al., 2018). The questionnaire also measures symptom severity for PTSD and cPTSD symptom clusters. It is the only self-report measure designed to diagnose ICD-11 cPTSD.
PTSD Checklist for the DSM-5 | Baseline (week 0), Treatment endpoint (week 12), Follow-up (3 months post treatment)
  The PTSD Checklist for the DSM-5 is a self-report measure used to assess the severity of PTSD symptoms as identified by the DSM-5 (American Psychiatric Association, 2013; Blevins et al., 2015). The measure is appropriate for evaluating treatment progress and changes in PTSD symptoms over time.
Biomarkers - Hormonal markers | Baseline (week 0), Treatment endpoint (week 12)
  Neurosteroid markers in the allopragnanolone pathway
Illness Intrusiveness Scale | Baseline (week 0), Treatment endpoint (week 12), Follow-up (3 months post treatment)
  The Illness Intrusiveness Scale is a 13-item self-report questionnaire assessing the impact of chronic illnesses such as mental illness on a person's daily life, functioning, and well-being (Fattori et al., 2016). The Illness Intrusiveness Scale covers three domains: relationships and personal development, instrumental life domains, and intimacy and leisure.
Biomarkers - Epigenetic | Baseline (week 0), Treatment endpoint (week 12)
  DNA methylation (epigenetic) markers: SLC6A4, which plays a crucial role in serotonin transportation; FKBP5, which is implicated in cortisol signalling; brain derived neurotrophic factor (BDNF), which supports neuronal growth, maturation, and maintenance; NR3C1, which codes for glucocorticoid receptors and regulates the HPA axis.
Biomarkers - Inflammatory | Baseline (week 0), Treatment endpoint (week 12)
  Inflammatory markers: CRP, which provides a proxy measurement for overall immune functioning; interleukin 6 (IL-6), a cytokine playing both pro- and anti-inflammatory roles; interferon-gamma (IFN-g), a pro-inflammatory cytokine; interleukin-10 (IL-10), an anti-inflammatory cytokine; tumor necrosis factor-alpha (TNF-a), another pro-inflammatory cytokine.

CONTACTS AND LOCATIONS:
Overall Officials: Benicio Frey, MD, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton; Sheryl Green, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton; Jenna Boyd, PhD, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided